CLINICAL TRIAL: NCT03843918
Title: A Phase I/II Study on the Safety and Efficacy of LAE001 in the Treatment of Metastatic Prostate Cancer
Brief Title: A Study on the Safety and Efficacy of LAE001 in the Treatment of Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This is phase I/II study, phase I study completed, phase II study started and enrolled 1 patient. Company strategy consideration to terminated phase 2 study finally.
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAE001CN2101
Record Dates: First submitted 2019-01-29; First posted 2019-02-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer Metastatic
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I: 3+3 design for dose escalation Phase II: designed as a single arm, multicenter trial
Masking Description: Phase I: Open label; Phase II: Open label;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LAE001+ADT (Experimental): LAE001+ADT
  Interventions: Drug: LAE001

INTERVENTIONS:
Drug: LAE001 — LAE001 BID will be orally administered until the subjects develop disease progression, intolerable adverse events, or trial withdrawal decided by the investigator/subject. The LAE001 dose adopted for the phase II study will be based on the RP2D determined in the phase I study.
  Other Names: CFG920

SUMMARY:
This study is a multicenter phase I/II study of the treatment of patients with metastatic prostate cancer. The objective of Phase I part is to study the safety and tolerability of LAE001 monotherapy in patients with metastatic castration-resistant prostate cancer, and determine the maximum tolerated dose (MTD) as well as the recommended phase II dose (RP2D) of the drug, the Phase II part is to assess the efficacy of LAE001 based on PSA in the treatment of patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
Phase I study of this study is a dose-escalating study with enrollment of patients with metastatic castration-resistant prostate cancer who have never received chemotherapy or who have received chemotherapy (chemotherapy failure or intolerance), and preferential enrollment of patients who had failed chemotherapy. The phase II study is a single arm, multicenter study based on ADT, and only patients with metastatic castration-resistant prostate cancer will be enrolled.

According to the results of a completed phase I dose-escalation trial and preclinical data on the drug, the initial dose proposed for this study is 50 mg BID, and one cycle will be 28 days. The escalated doses are 100 mg BID and 125 mg BID, two dose groups. If two or more cases of DLT occur for 100 mg BID, the dose may be reduced to 75 mg BID for investigation. If DLT occurs in two or more out of six patients for a certain dose group, the group with the dose preceding the testing dose will be determined to be the MTD dose group.

RP2D will be determined based on a comprehensive analysis of the safety, pharmacokinetic, pharmacodynamic and efficacy data of dose escalation. Where the MTD is determined, MTD is usually taken as the RP2D, or a dose lower than MTD is selected as the RP2D based on the combined data. If it is determined from the safety data that the dose can still be further increased, but the pharmacokinetic data indicate that the plasma concentration of LAE001 has reached steady-state saturation, the lowest dose that reaches steady-state saturation will be taken as the RP2D. According to the above principles, if the overall incidence of DLT at the dose is < 1/3, this testing dose will be determined as the RP2D. Six patients will be further enrolled and treated at the RP2D dose for sufficient pharmacokinetic data.

Phase II study is designed as a signle arm, multicenter trial on top of ADT therapy. Its primary objective is to assess the efficacy and safety of LAE001 in patients with metastatic castration-resistant prostate cancer. About 40 patients will be enrolled and assigned to the LAE001 treatment group on top of basic ADT therapy. Participant will be treated until the occurrence of disease progression (clinical evidence required), intolerance, judgement by the investigator that the patient is unsuitable to continue receiving treatment, death, or withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the trial procedures and content, and voluntarily signs the written informed consent form.
2. Male ≥ 18 years old.
3. Prostate adenocarcinoma as confirmed by histology or cytology, excluding neuroendocrine differentiation, signet ring cell carcinoma, and small cell carcinoma.
4. Evidence (such as bone scan or CT/MRI findings) of distant metastatic disease.
5. Phase I: According to the definition by PCWG3, disease progression after androgen deprivation therapy is as follows:

   • Disease progression, as defined by PCWG3, is the satisfaction of any of the following: According to elevations in PSA levels, there should be two consecutive elevations in PSA at least one week apart (if the third detected value is greater than the second detected value, the disease is determined to have progressed; if the third detected value is smaller than the second detected value, a fourth test is required to determine whether the PSA value is greater than the second detected value, and the interval between each test shall be at least one week), and the minimum value shall be equal to or greater than 1.0 ng/mL; PSA levels can be ignored for disease progression as assessed according to RECIST 1.1; progression of bone disease as defined by PCWG3, that is, the discovery of two or more new lesions via bone scan.

   • ECOG score of 0-1.

   • Dose-escalation phase: Patients with metastatic castration-resistant prostate cancer who have not received chemotherapy or who have received chemotherapy (chemotherapy failure or intolerance), with preferential enrollment of patients who had failed chemotherapy.

   Phase II: Patients with metastatic castration-resistant prostate cancer • ECOG score of 0-1.

   • Allow other previous treatment for mCRPC: Up to 1 cycle of palliative radiotherapy or surgical intervention to control the appearance of prostate cancer. Radiotherapy for the purpose of healing is not allowed. Radiation therapy must be completed at least 2 weeks before the first dose..
6. The subject underwent orchiectomy, or LHRH agonist or antagonist therapy before enrollment, and the therapy will be maintained throughout the entire study. The patient was at castration level during screening, i.e., his testosterone level was < 50 ng/dL or 1.7 nmol/L.
7. Adequate hematopoietic function:

   o White blood cell count, WBC ≥ 3,000/μL
   * Absolute neutrophil count, ANC ≥ 1,500/μL
   * Platelet count ≥ 100,000/μL
   * Hemoglobin ≥ 9 g/dL
8. Total serum bilirubin ≤ 1.5*ULN (total bilirubin ≤ 3*ULN, and direct bilirubin ≤ 1.5*ULN for patients known to have Gilbert syndrome).
9. AST (aspartate transaminase) and ALT (alanine transaminase) ≤ 2.5*ULN, and AST and ALT ≤ 5*ULN for patients with liver metastasis.
10. Serum creatinine ≤ 1.5*ULN.
11. Fasting plasma glucose ≤ 120 mg/dL or ≤ 6.7 mmol/L.(Appropriate treatment including insulin is accepted)
12. Normal levels of potassium, calcium and magnesium.

Exclusion Criteria:

1. Patients who had been treated with abiraterone acetate or enzalutamide.
2. Phase I: Patients who received anti-tumor therapy such as chemotherapy, radiotherapy, targeted therapy, and endocrine therapy with androgen receptor inhibitors within four weeks prior to the first dose (the time from the last treatment with nitrosourea or mitomycin chemotherapeutic agents is < 6 weeks, and the time from the last dose of bicalutamide or nilutamide is < 6 weeks).
3. Phase II: Patients who received any chemotherapy, radiotherapy or surgery for metastatic prostate cancer before randomization. Exceptions: ADT therapy (LHRH agonist or orchiectomy) before Day 1 of Cycle 1. Or >4 weeks since last use of bicalutamide or other generation antiandrogen receptor antagonist (please confirm with sponsor). Subjects may receive a course of palliative radiotherapy or surgery to treat symptoms caused by metastatic disease (e.g. spinal cord compression or obstruction), provided that it is administered at least 28 days prior to Day 1 of Cycle 1. All adverse events associated with such treatment must be alleviated to Grade 1 by Day 1 of Cycle 1.
4. Patients who underwent major surgery (major surgery refers to Grade 3 and Grade 4 surgery as defined in the "Administrative Measures for Clinical Application of Medical Technologies" promulgated on May 01, 2009) within 28 days before the study treatment, or who have not fully recovered from surgery (the investigator determines that the patient's participation in the clinical trial would pose a risk).
5. Patients with known severe cardiovascular diseases, including: myocardial infarction or thrombotic events in the past six months; unstable angina; heart failure of Class III or IV according to the criteria of the New York Heart Association (NYHA); QTc interval (QTcF) > 450 ms during the screening visit; G3 hypertension that cannot be controlled even with standard treatment, systolic blood pressure >160 mmHg or diastolic blood pressure>100 mmHg).
6. Patient who have not yet recovered from the toxicity of the former treatment regimen before drug administration on Day 1 of Cycle 1, and still have toxic reactions (excluding hair loss) above Grade 1 according to the grading scale of version 5.0 of the Common Terminology Criteria for Adverse Events (CTCAE).
7. Patients with clinically obvious gastrointestinal abnormalities that may affect the intake, transportation or absorption of drugs (such as patients who are unable to swallow, have chronic diarrhea or intestinal obstruction, or who had undergone total gastrectomy).
8. Patients with visceral metastasis involving the adrenal glands and central nervous system.
9. Patients with evidence of myelosuppression, and hydronephrosis in both kidneys as well as bladder neck obstruction that affects kidney function
10. Type I diabetes and type II diabetes that cannot be controlled by medication
11. Patients with a history of severe central nervous system diseases, including epilepsy.
12. Patients who had other malignant tumors (except for basal or squamous cell carcinoma) in addition to prostate cancer in the past five years, which are currently clinically significant and require intervention.
13. Patients who received 5α-reductase inhibitors (finasteride, dutasteride), estrogen, cyproterone and other drugs for treatment within four weeks before the first dose, and whose period of drug discontinuation has not exceeded five half-lives of the corresponding drugs; the drugs must have been discontinued for more than two weeks if the half-life is unknown.
14. Male patients whose sexual partners are women of childbearing age, where the patient and / or his sexual partner do not agree to use highly effective contraceptive measures (i.e. contraceptives with a low failure rate (less than or equivalent to 1% per year) when used consistently and correctly), and continued use of such measures until four weeks after drug discontinuation.
15. Patients who require systemic steroids or who had received systemic steroids (more than or equivalent to 10 mg of prednisone per day) 30 days before enrollment; topical, inhaled, ophthalmic or intra-articular medications are acceptable.
16. Patients who need to take diuretics (non-potassium-sparing).
17. Patients known to have pituitary or adrenal insufficiency.
18. Patients with known congenital or acquired immunodeficiency, active tuberculosis, etc.
19. Patients with active infection(s) that require systemic treatment within 10 days prior to signing the informed consent form.
20. Chronic hepatitis B carriers with untreated chronic active hepatitis B or with HBV DNA ≥ 1000 copies/mL (or ≥ 200 IU/mL), or patients with active hepatitis C.

21 The patient is currently receiving the following drugs and cannot discontinue the drugs at least one week before starting the study drug: Spironolactone Substrates of CYP1A2, CYP2E1 or CYP2C19, with a narrow therapeutic index Strong inhibitor or strong inducer of CYP1A2 Strong inhibitor of BSEP Grapefruit juice, and herbs such as St. John's wort, kava, ephedra, ginkgo biloba leaves, dehydroepiandrosterone, yohimbine, saw palmetto, and ginseng.

22. The patient is currently receiving a moderate or strong inhibitor or isoenzyme inducer of CYP3A. Patients taking strong inducers need to discontinue the drug for at least one week, and patients taking strong inhibitors need to at least discontinue the drug before receiving the study treatment.

23. Patients with other physical, psychological or social problems, including drug abuse, or who are deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT (Phase I) | up to 28 days
  To study the incidence of DLT in the first cycle of administration
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | through phase I part of study completion, an approximate average of 7 months
  To describe the incidence and severity of adverse events as assessed by CTCAE Version 5.0

SECONDARY OUTCOMES:
12-week PSA response rate | 12 weeks after randomization
  12-week PSA response rate Two consecutive measurements taken three to four weeks apart)
Overall response rate (ORR) | through study completion, an approximate average of 7 months
  Overall response rate (ORR) based on RECIST v1.1
Pharmacokinetic: Cmax | through phase I part of study completion, an approximate average of 7 months
  Collect plasma concentration of LAE001 at various time points and calculate Peak Plasma Concentration (Cmax)
Changes in Testosterone Levels | through phase I part of study completion, an approximate average of 7 months
  Observe changes in testosterone levels
Radiographic progression-free survival (rPFS) (Phase II) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, approximately up to 35 months
  Time from randomization to radiographic (as defined by Recist 1.1) progression or disease-induced death
PSA progression-free survival (Phase II) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, approximately up to 35 months
  Time from start of treatment to PSA progression
Overall response rate (ORR) (Phase II) | through phase II part of study completion, approximately up to 35 months
  Overall response rate (ORR) based on RECIST v1.1
12-month FFS rate (Phase II) | 12 months after randomization
  The rate of radiographic, clinical or PSA (as defined by PCWG3) progression or disease-induced death after 12 months treatment
Time to symptomatic skeletal event (SSE) (Phase II) | Time from the date of randomization to the date of documented symptomatic skeletal event,approximately up to 35 months
  Time to symptomatic skeletal event
Number of participants with adverse events as assessed by CTCAE v5.0 | through phase II part of study completion, approximately up to 35 months
  To describe the incidence and severity of adverse events as assessed by CTCAE Version 5.0
Pharmacokinetic: Tmax | through Phase I part of study completion, an approximate average of 7 months
  Collect plasma concentration of LAE001 at various time points and calculate Time to Peak Plasma Concentration (Tmax)
Pharmacokinetic: T 1/2 | through Phase I part of study completion, an approximate average of 7 months
  Collect plasma concentration of LAE001 at various time points and calculate half life
Pharmacokinetic: AUC0 - ∞ | through Phase I part of study completion, an approximate average of 7 months
  Collect plasma concentration of LAE001 at various time points and calculate Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic: CL | through Phase I part of study completion, an approximate average of 7 months
  Collect plasma concentration of LAE001 at various time points and calculate plasma clearance (CL)
Pharmacokinetic: Vd | through Phase I part of study completion, an approximate average of 7 months
  Collect plasma concentration of LAE001 at various time points and calculate volume of distribution
Changes in aldosterone levels | through phase I part of study completion, an approximate average of 7 months
  Observe changes in aldosterone levels
Changes in cortisol levels | through phase I part of study completion, an approximate average of 7 months
  Observe changes in cortisol levels
Changes in ACTH levels | through phase I part of study completion, an approximate average of 7 months
  Observe changes in ACTH levels

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD, Principal Investigator — Fudan University Shanghai Cnacer Center
Locations (2):
- China (2):
  - Fudan Cancer Hospital, Shanghai, Shanghai Municipality
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No